CLINICAL TRIAL: NCT05490017
Title: SYNERGY-1: A Phase 1 First-in-human, Randomized, Double Blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Escalating Single and Multiple Doses of KP104 in Healthy Subjects
Brief Title: To Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Escalating Single and Multiple Doses of KP104
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kira Pharmacenticals (US), LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KP104-101
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: KP104; Paroxysmal Nocturnal Hemoglobinuria; Single ascending Dose; Multiple Ascending Dose; First in Human; Complement Inhibitor; Healthy participants
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Part 1: Single Ascending Dose Cohort 1 (Experimental)
  Interventions: Drug: KP104
- Part 1: Single Ascending Dose Cohort 2 (Experimental)
  Interventions: Drug: KP104
- Part 1: Single Ascending Dose Cohort 3 (Experimental)
  Interventions: Drug: KP104
- Part 1: Single Ascending Dose Cohort 4 (Experimental)
  Interventions: Drug: KP104
- Part 1: Single Ascending Dose Cohort 5 (Experimental)
  Interventions: Drug: KP104
- Part 1: Single Ascending Dose Cohort 6 (Experimental)
  Interventions: Drug: KP104
- Part 1: Single Ascending Dose Cohort 7 (Experimental)
  Interventions: Drug: KP104
- Part 2: Multiple Ascending Dose Cohort 1 (Experimental)
  Interventions: Drug: KP104
- Part 2: Multiple Ascending Dose Cohort 2 (Experimental)
  Interventions: Drug: KP104
- Part 2: Multiple Ascending Dose Cohort 3 (Experimental)
  Interventions: Drug: KP104
- Part 1: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part 2: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KP104 — Participants will receive KP104 intravenous (IV) dose approximately for 1 hour or subcutaneous (SC) dose.
  Arms: Part 1: Single Ascending Dose Cohort 1; Part 1: Single Ascending Dose Cohort 2; Part 1: Single Ascending Dose Cohort 3; Part 1: Single Ascending Dose Cohort 4; Part 1: Single Ascending Dose Cohort 5; Part 1: Single Ascending Dose Cohort 6; Part 1: Single Ascending Dose Cohort 7; Part 2: Multiple Ascending Dose Cohort 1; Part 2: Multiple Ascending Dose Cohort 2; Part 2: Multiple Ascending Dose Cohort 3
Drug: Placebo — Participants will receive matching placebo which is KP104 vehicle containing sodium phosphate, sodium chloride, and L-Lysine Hydrochloride (L-Lys-HCL).
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, immunogenicity, pharmacokinetics, pharmacodynamics, and efficacy of KP104 in healthy volunteers. The study will be conducted in 2 parts: Part 1, the single ascending dose (SAD) is the first in human (FIH) study of KP104 and Part 2, multiple ascending dose (MAD).

ELIGIBILITY:
Inclusion Criteria:

* Weight of > 40 kilograms (kg) and < 120 kg at Screening.
* In good general health, determined by no clinically significant findings in the opinion of the Investigator from medical history, physical examination, 12-lead ECG, clinical laboratory findings, and vital signs at Screening and Check-in.
* Hemoglobin, hematocrit, white blood cell count, absolute neutrophil count, and platelet count results within the normal range at the Screening Visit; participants with Gilbert's disease with associated abnormalities of liver function tests are eligible for enrollment. Tests may be repeated at the discretion of the Investigator to confirm abnormalities.
* Creatinine clearance based on the Cockcroft-Gault equation of >= 80 milliliters per minute (ml/min).
* Females of childbearing potential and males must practice effective contraception from Screening until 28 days after the end of study (EOS) visit.
* Females of childbearing potential must have a negative pregnancy test at Screening and within 24 hours prior to dosing of study drug; for post-menopausal subjects, a blood sample will also be tested for follicle stimulating hormone to confirm post-menopausal status.

Exclusion Criteria:

* Any clinically significant underlying illness in the opinion of the Investigator.
* Any history or sign of significant chronic active or recurrent infection, or screening laboratory evidence consistent with a significant chronic active or recurrent infection requiring treatment with antibacterials, antivirals, or antifungals.
* Treatment of any infection with IV (within 30 days of Screening) or oral (within 14 days of Screening) antibacterials, antivirals, or antifungals.
* History of clinically significant hematologic or bone marrow disease or blood dyscrasias.
* History of meningococcal infection.
* History of tuberculosis.
* History of asplenia (functional or anatomical).
* Prior exposure to KP104.
* Known allergy to penicillin antibiotics or history of allergy or contraindication to required prophylactic antibiotic therapy to be used during the study.
* Known or suspected complement deficiency during screening.
* Positive serology for Hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV) at Screening.
* History of drug or alcohol abuse within 1 year of Screening in the opinion of the investigator, or a positive test for drugs of abuse or alcohol at Screening or Check-in.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting Treatment Emergent Adverse Events (TEAEs) | Up to Day 85
  An Adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding), symptom, or disease or any worsening of a pre-existing condition temporally associated with the use of a study drug, whether or not related to study drug. A TEAE is defined as any AE that started or worsened in severity on or after the first dose of study treatment.
Number of participants reporting Treatment Emergent Serious Adverse Events (TESAEs) | Up to Day 85
  A TESAE is defined as any AE that started or worsened in severity on or after the first dose of study treatment.
Number of participants with Dose-limiting toxicities (DLT) | Up to Day 85
  A DLT is defined as any adverse event considered by the investigator to be KP104-related with a severity greater than or equal to (>=) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grade 3 which also represents a shift from baseline clinical status of > 1 NCI CTCAE grade. A hypersensitivity/administration reaction occurring with a severity of Grade 2 despite the use of pre-medications will also be designated as a DLT.
Number of participants reporting AEs of Special interests (AESIs) | Up to Day 85
  An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease or any worsening of a pre-existing condition temporally associated with the use of a study drug, whether or not related to study drug. Number of participants with AESIs including infections and local or systemic administration reactions will be assessed.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of KP104 | Up to Day 29
Area under the concentration-time profile (AUC) of KP104 | Up to Day 29
Change from baseline in total and free serum C5 levels | Baseline and up to Day 29
Change from baseline in rabbit red blood cell (RBC) assay | Baseline and up to Day 29

OTHER OUTCOMES:
Changes in serum free C5 levels to Minimum concentration (Cmin) correlation | Baseline and up to Day 29
Changes in serum free C5 levels to AUC correlation | Baseline and up to Day 29
Changes in C3b activity to Cmax correlation | Baseline and up to Day 29
Changes in C3b activity to Cmin correlation | Baseline and up to Day 29
Changes in C3b activity to AUC correlation | Baseline and up to Day 29
Changes in rabbit RBC lysis to Cmax correlation | Baseline and up to Day 29
Changes in rabbit RBC lysis to Cmin correlation | Baseline and up to Day 29
Changes in rabbit RBC lysis to AUC correlation | Baseline and up to Day 29
Immunogenicity of KP104 | Up to Day 29
Maximum tolerated dose (MTD) of KP104 | Up to Day 29
Optimal biologic dose (OBD) of KP104 | Up to Day 29
Number of participants with clinically significant changes in laboratory values, electrocardiograms (ECGs), physical examinations, and vital signs | Up to Day 29
Changes in serum free complement component C5 levels to Cmax correlation | Baseline and up to Day 29
Dose optimization of KP104 | Up to Day 29
Systemic clearance (Cl) of KP104 | Up to Day 29
Elimination half-life (t½) of KP104 | Up to Day 29
Change from baseline in complement component of C3b activity assay | Baseline and up to Day 29
Absolute bioavailability of KP104 administered SC (F) | Up to Day 29
Change from baseline in Factor H (FH) serum levels | Baseline and up to Day 29

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: Yes